CLINICAL TRIAL: NCT05940883
Title: A 2-Part, Randomized, Phase I Study to Evaluate the Pharmacokinetics,Safety and Tolerability of Y-2 Sublingual Tablet in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics,Safety and Tolerability of Y-2 Sublingual Tablet in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0308-Y-2-101
Record Dates: First submitted 2023-06-27; First posted 2023-07-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Y-2 sublingual tablet dose group 1 (Experimental)
  Interventions: Drug: Y-2 Sublingual Tablet
- Y-2 sublingual tablet dose Group 2 (Experimental)
  Interventions: Drug: Y-2 Sublingual Tablet
- Y-2 sublingual tablet dose Group 3 (Experimental)
  Interventions: Drug: Y-2 Sublingual Tablet
- Y-2 sublingual tablet dose Group 4 (Experimental)
  Interventions: Drug: Y-2 Sublingual Tablet
- Y-2 sublingual tablet dose Group 5 (Experimental)
  Interventions: Drug: Y-2 Sublingual Tablet
- Placebo (Placebo Comparator): Certain subjects in group 1 and group 2 will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Y-2 Sublingual Tablet — Subjects will receive one Y-2 sublingual tablet sublingually once daily for Day1 and Day 19 and twice daily for Day 6 to Day 18.
  Arms: Y-2 sublingual tablet dose group 1
Drug: Y-2 Sublingual Tablet — Subjects will receive two Y-2 sublingual tablets sublingually once daily for Day1 and Day 19 and twice daily for Day 6 to Day 18.
  Arms: Y-2 sublingual tablet dose Group 2
Drug: Y-2 Sublingual Tablet — Subjects will receive Y-2 sublingual tablet with 3 different conditions once daily for Day1 Day 6 and Day 11. Day 1 with condition A, Day 6 with condition B and Day 11 with condition C.
  Arms: Y-2 sublingual tablet dose Group 3
Drug: Y-2 Sublingual Tablet — Subjects will receive Y-2 sublingual tablet with 3 different conditions once daily for Day1 Day 6 and Day 11. Day 1 with condition B, Day 6 with condition C and Day 11 with condition A.
  Arms: Y-2 sublingual tablet dose Group 4
Drug: Y-2 Sublingual Tablet — Subjects will receive Y-2 sublingual tablet with 3 different conditions once daily for Day1 Day 6 and Day 11. Day 1 with condition C, Day 6 with condition A and Day 11 with condition B.
  Arms: Y-2 sublingual tablet dose Group 5
Drug: Placebo — Placebo, sublingually, single and multiple ascending dosing in group 1 and 2 subjects.
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics(PK) of Y-2 sublingual tablet in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
  2. Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 and weight ≥ 50kg at screening.
  3. A condition of general good health, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
  4. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following condition applies:

     * Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 Contraceptive Guidance, OR
     * A WOCBP who agrees to follow the contraceptive guidance in Appendix 1 Contraceptive Guidance from screening through at least 90 days after the last dose of study drug; a WOCBP must have a negative beta-human chorionic gonadotropin (β-hCG) test at screening and baseline prior to administration of investigational product.

Exclusion Criteria:

1. Subject has a history of any clinically significant cardiac, respiratory (including asthma, bronchospasm), renal, hepatic,gastrointestinal, psychiatric, neurologic, hematologic or rheumatic disease, or psychiatric disease or disorder, current acute or chronic infections, or other abnormality that may affect safety, or potentially influence the study results, judged by the investigator or designee.
2. Evidence or history of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma.
3. Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 90 days or 5 half-lives (whichever is longer) prior to Day 1.
4. Receipt of any investigational product within 30 days or 5 halflives (whichever is longer) prior to Day 1.
5. Will have vaccination with live virus, attenuated live virus, or any live viral components within the 30 days prior to Day 1 or is to receive these vaccines at any time during study period or within 90 days after last dose.
6. Female subject who is pregnant, breastfeeding or is considering becoming pregnant during the study or for approximately 90 days after the last dose of study drug.
7. Male subject who is considering fathering a child or donating sperm during the study or for approximately 90 days after the last dose of study drug.
8. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to enroll this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events（Part 1) | Until follow-up（Day26）or early termination
  To evaluate the safety and tolerability following single and multiple administrations of Y-2 sublingual tablet in healthy adult subjects in part 1.
Maximum concentration（Cmax）in Part 2 healthy adult subjects | Day1，Day2， Day6，Day7，Day11，Day12
  To evaluate the effects of different administration conditions on the PK of edaravone and dexborneol in plasma following single administration of Y-2 sublingual tablet in healthy adult subjects in part 2.
Time for Cmax (Tmax) in Part 2 healthy adult subjects | Day1，Day2， Day6，Day7，Day11，Day12
  To evaluate the effects of different administration conditions on the PK of edaravone and dexborneol in plasma following single administration of Y-2 sublingual tablet in healthy adult subjects in part 2.
Area under the curve (AUC) in Part 2 healthy adult subjects | Day1，Day2， Day6，Day7，Day11，Day12
  To evaluate the effects of different administration conditions on the PK of edaravone and dexborneol in plasma following single administration of Y-2 sublingual tablet in healthy adult subjects in part 2.
Terminal elimination half-life（t1/2） in Part 2 healthy adult subjects | Day1，Day2， Day6，Day7，Day11，Day12
  To evaluate the effects of different administration conditions on the PK of edaravone and dexborneol in plasma following single administration of Y-2 sublingual tablet in healthy adult subjects in part 2.

SECONDARY OUTCOMES:
Maximum concentration（Cmax）in Part 1 healthy adult subjects | Day1，Day2，Day6 and Day18 to Day20
  To characterize the PK of edaravone and dexborneol in plasma following single and multiple administrations of Y-2 sublingual tablet in healthy adult subjects in part 1.
Time for Cmax (Tmax) in Part 1 healthy adult subjects | Day1，Day2，Day6 and Day18 to Day20
  To characterize the PK of edaravone and dexborneol in plasma following single and multiple administrations of Y-2 sublingual tablet in healthy adult subjects in part 1.
Area under the curve (AUC) in Part 1 healthy adult subjects | Day1，Day2，Day6 and Day18 to Day20
  To characterize the PK of edaravone and dexborneol in plasma following single and multiple administrations of Y-2 sublingual tablet in healthy adult subjects in part 1.
Terminal elimination half-lifet（1/2 ）in Part 1 healthy adult subjects | Day1，Day2，Day6 and Day18 to Day20
  To characterize the PK of edaravone and dexborneol in plasma following single and multiple administrations of Y-2 sublingual tablet in healthy adult subjects in part 1.
Adverse Events（Part 2) | Until follow-up（Day18）or early termination
  To evaluate the safety following different single administration conditions of Y-2 sublingual tablet in healthy adult subjects in part 2.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, MD, Principal Investigator — Parexel
Locations (1):
- Parexel International Los Angeles Early Phase Clinical Unit, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No